CLINICAL TRIAL: NCT04869241
Title: Changes in Muscle Activation of Serratus Anterior, Deltoid (Anterior) and Trapezius (Upper and Lower) According to the Methods of Carrying Backpacks
Brief Title: Changes in Muscle Activation When Carrying Backpacks
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of a principal investigator
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Director, Bundang CHA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BundangCHA
Record Dates: First submitted 2021-04-08; First posted 2021-05-03 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Shoulder Muscle Activation; Surface Emg
Keywords: backpack; shoulder muscle activation; surface emg; deltoid, serratus anterior, trapezius
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Group measuring shoulder muscle activities by surface EMG with carrying backpacks forward
  Interventions: Diagnostic Test: surface EMG

INTERVENTIONS:
Diagnostic Test: surface EMG — Carrying backpacks forward or backward

SUMMARY:
To investigate change of shoulder muscles by measuring muscle activity according to the position of the backpack.

DETAILED DESCRIPTION:
Most of modern people, including students and office workers, wear backpacks for a considerable amount of time. There have been prior studies on the change in muscle activity around the spine and shoulders muscles according to the weight of the backpack, but studies on the change in muscle activity according to the direction of the bag are insufficient. So this study is to evaluate the effect on the musculoskeletal system by comparing the activity of the muscles around the shoulder according to the anterior or posterior wearing of the backpack.

Muscles around the shoulder are composed of: Serratus anterior, trapezius(upper and lower) which control scapular movement and deltoid muscles which activate shoulder abduction directly. We would like to focus change of these muscles's activities when carrying a backpack according to the anterior or posterior direction and bilateral or unilateral.

To measure muscle activity, eight-channel electromyography (EMG) Using Nicolet EDX (Natus Medical Inc., San Carolos, CA, USA), surface EMG (sEMG) signal were used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults from 20s to 50s

Exclusion Criteria:

* Restriction of joint motion range of shoulder and elbow
* Hisory of upper limb surgery in the past 6 months
* If there is an external wire such as a temporary external pacemaker or central line guide wire

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Root mean square of each muscle activation | through study completion, an average of 1 year
  Quantification of muscle activity

CONTACTS AND LOCATIONS:
Overall Officials: Kyunghoon Min, MD, PhD, Study Director — Department of Rehabilitation Medicine, CHA Bundang Medical Center, CHA University School of Medicine
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes